CLINICAL TRIAL: NCT05393583
Title: In-hospital Versus DAy Care Hysterectomy in Transgender Men
Acronym: IDAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EC/2018/1387
Record Dates: First submitted 2022-01-21; First posted 2022-05-26 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Outpatient Hysterectomy in Transmen

STUDY DESIGN:
Intervention Model Description: 2-armed study
  * arm 1: outpatient hysterectomy (discharge the day of the operation)
  * arm 2: inpatient hysterectomy (1 night hospital stay)
Masking Description: Blinding not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient (Experimental): Discharge on the day of hysterectomy
  Interventions: Procedure: Outpatient hysterectomy
- Inpatient (Active Comparator): Discharge after 1 night stay in the hospital
  Interventions: Procedure: Inpatient hysterectomy

INTERVENTIONS:
Procedure: Outpatient hysterectomy — Discharge on the day of the hysterectomy
  Arms: Outpatient
Procedure: Inpatient hysterectomy — 1 night hospital stay after hysterectomy
  Arms: Inpatient

SUMMARY:
In this trial 2 groups of transmen who are getting a hysterectomy will be compared: inpatient vs outpatient.

DETAILED DESCRIPTION:
In this trial transmen who consultate for a hysterectomy are randomised over 2 groups: inpatient vs outpatient.

In the inpatient group the participant stays 1 night in the hospital after the laparoscopic hysterectomy. The outpatient group can leave the hospital the day of the operation. Standard care after laparoscopic hysterectomy is 2 nights hospital stay.

Through this trial the investigators would like to answer following questions:

* Is hysterectomy in dayclinic as safe as a hysterectomy in an outpatient setting?
* Is there a higher complication/re-admission rate with hysterectomy in outpatient setting?
* Are patients as satisfied with the length of hospital stay in an inpatient hysterectomy?
* Is the need for pain medication higher in the inpatient group? Do this patients experience more postoperative pain?
* Is there a loss in 'quality of life' with hysterectomy in inpatient setting?
* Are patients who have the hysterectomy in dayclinic more anxious/worried?

The primary objective is the satisfaction of the patient with the length of hospital stay. The other indicators will be seen as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* transgender man
* 18y or older
* registers for a total hysterectomy at the genderclinic of UZ Gent.

Exclusion Criteria:

* simultaneous planned breast surgery/scar corrections
* ASA score 3-4
* persons with mental retardation or severe psychiatric disorder
* persons without an adult caretaker / partner present the first night after discharge from the hospital

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — transmen
Enrollment: 104 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the length of hospital stay after 1 week assessed by the VAS (visual analogue scale) | Day 7
  Satisfaction of the patient with the length of hospital stay 1 week after surgery assessed by a Visual Analogue Scale ranging from 0 to 100 (with 100 being extremely satisfied)
Satisfaction with the length of hospital stay after 6 weeks assessed by the VAS (visual analogue scale) | Day 42
  Satisfaction of the patient with the length of hospital stay 6 weeks after surgery assessed by a Visual Analogue Scale ranging from 0 to 100 (with 100 being extremely satisfied)

SECONDARY OUTCOMES:
Pain scores | Day 0 to 7
  Pain will be measured by using a Visual Analogue Scale for pain ranging from 0 to 10 (with 10 being the worst pain ever)
Analgesics use | Day 0 to 7
  The amount of analgesics used every day
Type and number of intra-operative complications | Day 0
Type and number of postoperative complications | Day 42
Readmission rate | Day 42
Postoperative quality of recovery (QoR)-15 score | Day 1, day 2 and day 42
  The QoR-15 is a patient-reported outcome questionnaire that measures the quality of recovery after surgery and anaesthesia. Each question is scored from 0 (= "none of the time") to 10 (= "all of the time") for positive items; for negative items the scoring is reversed (maximum score 150).
Postoperative wellbeing through the Hospital Anxiety and Depression Scale (HADS) | Day 1, day 2 and day 42
  Postoperative wellbeing will be assessed by using the HADS. The HADS is a 14-question instrument that measures anxiety and depression. Each question is scored between 0 (no impairment) and 3 (severe impairment), with a maximum score of 21 for anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dedden SJ, Geomini PMAJ, Huirne JAF, Bongers MY. Vaginal and Laparoscopic hysterectomy as an outpatient procedure: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2017 Sep;216:212-223. doi: 10.1016/j.ejogrb.2017.07.015. Epub 2017 Jul 22. PMID 28810192
- [Background] Kisic-Trope J, Qvigstad E, Ballard K. A randomized trial of day-case vs inpatient laparoscopic supracervical hysterectomy. Am J Obstet Gynecol. 2011 Apr;204(4):307.e1-8. doi: 10.1016/j.ajog.2010.11.014. Epub 2011 Jan 26. PMID 21272844
- [Derived] Verberckmoes B, van Wessel S, Hamerlynck T, Bosteels J, Coppens M, Weyers S. Ambulatory Versus Inpatient Total Laparoscopic Hysterectomy in Trans Men: A Randomised Controlled Non-Inferiority Trial. BJOG. 2026 Jan;133(1):52-60. doi: 10.1111/1471-0528.18340. Epub 2025 Aug 26. PMID 40856135